CLINICAL TRIAL: NCT03654872
Title: Clostridium Difficile Virulence Mechanism Study by Collecting Stool Samples From Clostridium Difficile Infection Patients (CDVM Study)
Brief Title: Clostridium Difficile Virulence Mechanism Study (CDVM Study)
Acronym: CDVM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Sunny Wong, Principal Investigator, Clinical Assistant Professor, Chinese University of Hong Kong
Other Study IDs: CDVMProtocol
Record Dates: First submitted 2018-08-19; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Clostridium Difficile Infection; Clostridium Difficile
Keywords: ribotypes; Hong Kong; virulence mechanism
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — DNA from stool maybe extracted for analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is an observational study to collect stool samples from patients with Clostridium difficile infection (CDI) to investigate the virulence mechanisms of C. difficile ribotypes in Hong Kong, mainly ribotype 002. No intervention is involved.

DETAILED DESCRIPTION:
This is an observational study to collect stool samples from patients with Clostridium difficile infection (CDI), aims to (1) to investigate the virulence mechanisms of C. difficile ribotype 002, by analysing its growth, cytotoxicity, and metabolite production in vitro and in vivo. The investigators also aim (2) to compare these virulence mechanisms with other common ribotypes in Asia, and (3) to correlate these with important clinical outcomes. The results of this study will have a major significance to the medical and scientific community. The results of this study will have a major significance to the medical and scientific community. The mechanistic data will point to important molecular pathways that can be targeted for novel therapies; whereas the phenotypic data will inform the investigators of its virulence and therefore will be useful for disease surveillance and public health interventions. The identified toxin(s) and metabolite(s) may be useful as prognostic biomarkers to stratify patients with different outcomes, as patients with a worse outcome may require more aggressive therapy. Given the prevalence and severity of this ribotype, the results will be useful for gastroenterologists, microbiologists, infectious diseases physicians and public health specialists in the Asia Pacific region.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of CDI, as documented by diarrheal symptoms and positive stool test result for C. difficile toxin or toxigenic C. difficile, or colonoscopic findings of pseudomembranous colitis (PMC).
* Patients aged over or equal to 18 years old.
* Patients able and willing to provide informed consent.

Exclusion Criteria:

* Patients with concomitant infection by other microbes such as Salmonella, Campylobacter, Vibrio, Shigella, and Escherichia coli.
* Patients under 18 years old.
* Patients who cannot give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects will be identified and recruited under the suitable patients pool in the apply site. If the subjects are confirmed to have diarrheal symptoms and positivie stool result of Clostridium difficile, the subjects will be recruited in the wards and will only be recruited if they sign the informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 227 (Estimated)
Dates: Start 2018-06-30 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Isolate Clostridium difficile from patients' stool for ribotyping to identify which ribotype was the Clostridium difficile from the patient. | 1 year
  Clostridium difficile will be isolated from stool sample of the patients and will be used for ribotyping. Ribotyping will be done to the Clostridium difficile strain isolated to classify them into different ribotypes. This is to measure the number of patients with a particular ribotype. Virulence mechanism will also be evaluated through experiments with isolated bacteria on growth curve, toxin production, sporulation, germination and adhesion.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sunny Wong, Principal Investigator — Institute of Digestive Disease, Department of Medicine and Therapeutics, Faculty of Medicine, The Chinese University of Hong Kong, Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT03654872/Prot_000.pdf